CLINICAL TRIAL: NCT02286869
Title: Cardioventilatory Coupling in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Fatebenefratelli Sacco (Other)
Collaborators: Tommaso Fossali (Other); Stefano Guzzetti (Unknown); Andrea Marchi (Unknown); Alberto Porta (Unknown); Beatrice Borghi (Unknown)
Responsible Party: Principal Investigator, Riccardo Colombo, Cardioventilatory coupling in critically ill, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CaVeCo
Record Dates: First submitted 2014-11-04; First posted 2014-11-10 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Critically Ill
Keywords: mechanical ventilation; autonomic nervous system; heart rate variability; cardioventilatory coupling
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pressure Controlled Ventilation (Experimental): INTERVENTION: respiratory trial in pressure controlled mode: (i) the inspiratory pressure is set up to obtain the same tidal volume than baseline, (ii) the imposed respiratory rate is the same respiratory rate than baseline.
  The positive end expiratory pressure and fractional inspiratory oxygen are unchanged from the baseline.
  After an acclimation period of 10 min, electrocardiographic, arterial pressure and respiratory waves are recorded for 30 min.
  Interventions: Procedure: Three different mechanical ventilation modes
- Pressure Support Ventilation (Experimental): INTERVENTION: respiratory trial in pressure support mode: (i) the inspiratory pressure is set up to obtain the same tidal volume than baseline, (ii) the inspiratory trigger is a flow-trigger with medium sensitivity.
  The positive end expiratory pressure and fractional inspiratory oxygen are unchanged from the baseline. In this ventilatory mode the respiratory rate is not imposed because is driven by the patient's respiratory effort.
  After an acclimation period of 10 min, electrocardiographic, arterial pressure and respiratory waves are recorded for 30 min.
  Interventions: Procedure: Three different mechanical ventilation modes
- Neurally Adjusted Ventilatory Assist (Experimental): INTERVENTION: respiratory trial in Neurally Adjusted Ventilatory Assist (NAVA) mode: (i) NAVA-level (gain) is set up to obtain the same tidal volume than baseline, (ii) the inspiratory trigger is a neural trigger set at 0.5 microVolt.
  The positive end expiratory pressure and fractional inspiratory oxygen are unchanged from the baseline. In this ventilatory mode the respiratory rate is not imposed because is driven by the patient's respiratory effort.
  After an acclimation period of 10 min, electrocardiographic, arterial pressure and respiratory waves are recorded for 30 min.
  Interventions: Procedure: Three different mechanical ventilation modes

INTERVENTIONS:
Procedure: Three different mechanical ventilation modes — patients are randomly assigned to every arm. Baseline is the period immediatly before the study phase. The study phase is the sequence of three consecutive trials of different modes of mechanical ventilation. Every trial lasts 30 min plus 10 min of acclimation.

SUMMARY:
This study measures the cardioventilatory coupling in critically ill patients during mechanical ventilation in controlled mode (pressure controlled) and in patient-driven mode (pressure support and neurally adjusted ventilatory assist).

DETAILED DESCRIPTION:
Intrathoracic pressure oscillations due to positive pressure ventilation induce cyclic modifications of activity of the pulmonary vascular receptors and cardiac mechanoceptors. These effects changes the autonomic nervous system modulation with modification of both sympathetic and vagal activity.

Cardio-ventilatory interaction recently has been studied through the heart rate variability in critically ill mechanical ventilated patients. The analysis of the power spectrum density provides information about the power (the variance of beat-to-beat interval) is distributed as frequencies' function. Healthy spontaneously breathing subjects show a cyclic inspiratory increase and expiratory decrease of heart rate, and 'phase coupling' between heart beats and respiration (causing heart beats to occur at constant phases of the respiratory cycle), commonly known as cardioventilatory coupling. These phenomena originate from a complex interplay of several mechanisms including central drive, feedback from arterial baroreceptors, feedback from thoracic and lung stretch receptors, and non-neural mechanisms intrinsic to the heart, which are not fully understood. Although the physiological importance of respiratory sinus arrhythmia and cardioventilatory coupling have not been elucidated, several authors suggested that they might improve ventilation/perfusion matching through a redistribution of heart beats (and consequently of perfusion) within the respiratory cycle, with beneficial effects on gas exchange. Furthermore, decreased respiratory sinus arrhythmia amplitude has been used as an indicator of impaired autonomic control and of poor clinical outcome, also during mechanical ventilation.It has been shown that during controlled mechanical ventilation the respiratory sinus arrhythmia amplitude is considerably reduced and the cardioventilatory coupling generally abolished. Theoretically, mechanical ventilation modes that assist the respiratory pump upon triggering by the patient, such as pressure support ventilation (PSV) might maintain higher respiratory sinus arrhythmia levels through centrally-originated phasic vagal modulation compared to controlled mechanical ventilation. In addition, mechanical ventilation with breath-by-breath variable tidal volumes, so-called 'variable ventilation', could better preserve respiratory sinus arrhythmia and cardioventilatory coupling, and this might play a role in the improved arterial oxygenation found in different models of acute lung injury, although with variable results, when comparing variable and conventional mechanical ventilation. In anesthetized experimental animals the cardioventilatory coupling was more preserved during pressure assisted ventilation than pressure controlled ventilation. If these findings could be present in the humans is yet unknown. Furthermore, it has been demonstrated that some new methodologies of assisted ventilation, such as the neurally adjusted ventilatory assist (NAVA), increase the breath-to-breath variability and tidal volume variability, but their effects on cardioventilatory coupling are not understood.

The study aims to measure the heart rate variability, the respiratory rate variability and the cardioventilatory coupling in critically ill patients during mechanical ventilation both in controlled mode (pressure controlled) and in assisted mode (pressure support ventilation and NAVA).

Methods enrolled patients are connected to a S/5 ICU monitor (GE, Helsinki, Finland) and are mechanically ventilated with a Servo-I ventilator (Maquet, Germany) provided with diaphragmatic electrical activity module (EAdi, Maquet, Germany). A nasogastric 16-Fr EAdi catheter is positioned in all patients. A sequence of three consecutive study phases of different mechanical ventilation modes (PCV, PSV, and NAVA) is started. The sequence of ventilatory modes is randomized for every patient. After a 10 min acclimation period for each study phase, electrocardiographic, arterial pressure and ventilatory waves are collected for consecutive 30 min to a laptop pc via S/5 Collect (GE, Helsinki, Finland) and NAVA Tracker (Maquet, Germany) software for Windows.

Heart rate variability analysis Linear analysis Sequences of 300 consecutives heart beats are selected inside each experimental phase. The mean and the variance of heart period are expressed in msec and msec^2 respectively. Autoregressive spectral density is factorized into components each of them characterized by a central frequency. A spectral component is labeled as LF if its central frequency is between 0.04 and 0.15 Hz, while it is classified as HF if its central frequency is between 0.15 and 0.5 Hz. The HF power is considered to represent respiration-driven vagal modulation of heart rate. To rule out the effect of changes of total power spectrum densities on LF and HF components, spectral values are also expressed in normalized units (NU). Normalization consisted in dividing the power of a given spectral component by the total power minus the power below 0.04 Hz (Very Low Frequency [VLF] spectral component), and multiplying the ratio by 100. The ratio of the LF power to the HF (LF/HF) is considered an indicator of the balance between sympathetic and vagal modulation directed to the heart.

Nonlinear analysis Non-linear analysis was conducted by means of symbolic analysis. The symbolic analysis is conducted on the same sequences of 300 consecutive heart beats that are used for the autoregressive analysis. The whole range of the R-to-R interval into each series is uniformly divided in 6 slices (symbols) and pattern of 3 consecutive heart beat intervals were considered. Thus each sequence of 300 heart beats had its own R-to-R range and 298 consecutive triplets of symbols. The Shannon entropy of the distribution of the patterns is calculated to provide a quantification of the complexity of the pattern distribution. All triplets of symbols are grouped into 3 possible patterns of variation: (i) no variation (0V, all 3 symbols were equal), (ii) 1 variation (1V, 2 consequent symbols were equal and the remaining symbol was different), (iii) patterns with 2 variations (2V, all symbols were different from the previous one). Previously, the percentage of 0V patterns was found to increase (and 2V decrease) in response to sympathetic stimuli, whereas 2V patterns increased (and 0V decreased) in response to vagal stimuli. The percentage of the patterns 0V and 2V was calculated, and the 0V/2V ratio was calculated to estimate the balance between sympathetic and vagal modulation.

Cardioventilatory coupling analysis Phase synchronization method for quantification of coupling between weakly coupled self-sustained oscillators (here heart and ventilator) will be implemented. The idea behind is that a good ventilatory mode should produce cardio-respiratory coordination indistinguishable from that observed in healthy subject during spontaneous breathing at the same frequency and amplitude. Phase synchronization technique is complemented with joint symbolic analysis and cross-conditional entropy assessing of cardio-respiratory coupling in terms of degree of repeatability of coordination schemes between heart rate signal and ventilation. These approaches have the main advantages that they are less sensitive to non-stationarities and they are capable of capturing nonlinear couplings over shorter data sequences.

Sample size given a heart rate variability total variance equal to 1000 msec^2, to detect a difference of 300 msec^2 (with a standard deviation of 200 msec^2) between the study phases with an alpha error=0.05, power=80%, effect size=0.4, 22 patients will be recruited.

The normal distribution is checked with Kolmogorov-Smirnov test. Two tails Student t test for dependent or independent sample as needed, or Wilcoxon- U test in case of not normal distribution are employed. Repeated measures are analyzed with one way analysis of variance (ANOVA) followed by post-hoc Bonferroni's test.

ELIGIBILITY:
Inclusion Criteria:

patients consecutively admitted to the mixed intensive care unit of the Luigi Sacco Hospital with (all the following):

* mechanical ventilation with an expected duration ≥ 48 hours
* acute respiratory failure due to ALI/ARDS or COPD exacerbation or pneumonia or severe sepsis/septic shock
* age between 18 and 75 years old

Exclusion Criteria:

* contraindications to esophageal tube positioning (i.e. esophageal varices, bleeding from upper enteric tract in the past 30 days)
* history of esophageal or gastric or thoracic surgery
* history of neuromuscular disease or stroke or head trauma
* history of thyroidal or adrenal dysfunction
* positive end expiratory pressure ≥ 10 cmH2O and/or inspiratory oxygen fraction ≥ 0.60, or intrinsic positive end expiratory pressure ≥ 8 cmH2O
* needing for neuromuscular blocking drugs administration
* patients unable to undergo to patient-driven mechanical ventilation mode (i.e. coma, excessive sedation)
* mechanical circulatory support (i.e. intra-aortic balloon, extracorporeal membrane oxygenation)
* norepinephrine ≥0.3 mcg/kg/min or epinephrine ≥0.05 mcg/kg/min or dobutamine ≥2.5 mcg/kg/min
* non sinus cardiac rhythm or ectopic beats exceeding ≥5% of normal sinus beats
* acute or chronic heart failure with reduced or preserved ejection fraction
* recent acute miocardial infarct ≤6 months
* recent recovery from respiratory failure or pneumonia or severe sepsis/septic shock ≤30 days
* therapy with beta-blockers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
to measure the cardioventilatory coupling in mechanically ventilated critically ill patients during three different mechanical ventilation settings | 120 min
  to measure the cardioventilatory coupling in mechanically ventilated critically ill patients during three different modes of mechanical ventilation: (i) Pressure Controlled Ventilation, (ii)

SECONDARY OUTCOMES:
to measure the heart rate variability in mechanically ventilated critically ill patients during three different mechanical ventilation settings | 120 min
  to measure the heart rate variability in mechanically ventilated critically ill patients during three different modes of mechanical ventilation: (i) Pressure Controlled Ventilation, (ii)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Luigi Sacco Hospital, Milan
  - Istituto Clinico Humanitas, Rozzano

REFERENCES:
- [Background] Pagani M, Lombardi F, Guzzetti S, Rimoldi O, Furlan R, Pizzinelli P, Sandrone G, Malfatto G, Dell'Orto S, Piccaluga E, et al. Power spectral analysis of heart rate and arterial pressure variabilities as a marker of sympatho-vagal interaction in man and conscious dog. Circ Res. 1986 Aug;59(2):178-93. doi: 10.1161/01.res.59.2.178. PMID 2874900
- [Background] Nollo G, Faes L, Porta A, Antolini R, Ravelli F. Exploring directionality in spontaneous heart period and systolic pressure variability interactions in humans: implications in the evaluation of baroreflex gain. Am J Physiol Heart Circ Physiol. 2005 Apr;288(4):H1777-85. doi: 10.1152/ajpheart.00594.2004. Epub 2004 Dec 16. PMID 15604132
- [Background] Rosenblum MG, Cimponeriu L, Bezerianos A, Patzak A, Mrowka R. Identification of coupling direction: application to cardiorespiratory interaction. Phys Rev E Stat Nonlin Soft Matter Phys. 2002 Apr;65(4 Pt 1):041909. doi: 10.1103/PhysRevE.65.041909. Epub 2002 Mar 28. PMID 12005875
- [Background] Porta A, Baselli G, Lombardi F, Montano N, Malliani A, Cerutti S. Conditional entropy approach for the evaluation of the coupling strength. Biol Cybern. 1999 Aug;81(2):119-29. doi: 10.1007/s004220050549. PMID 10481240
- [Background] Porta A, Guzzetti S, Montano N, Furlan R, Pagani M, Malliani A, Cerutti S. Entropy, entropy rate, and pattern classification as tools to typify complexity in short heart period variability series. IEEE Trans Biomed Eng. 2001 Nov;48(11):1282-91. doi: 10.1109/10.959324. PMID 11686627
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Galletly DC, Larsen PD. Inspiratory timing during anaesthesia: a model of cardioventilatory coupling. Br J Anaesth. 2001 Jun;86(6):777-88. doi: 10.1093/bja/86.6.777. PMID 11573583
- [Background] Giardino ND, Glenny RW, Borson S, Chan L. Respiratory sinus arrhythmia is associated with efficiency of pulmonary gas exchange in healthy humans. Am J Physiol Heart Circ Physiol. 2003 May;284(5):H1585-91. doi: 10.1152/ajpheart.00893.2002. Epub 2003 Jan 23. PMID 12543637
- [Background] Hayano J, Yasuma F, Okada A, Mukai S, Fujinami T. Respiratory sinus arrhythmia. A phenomenon improving pulmonary gas exchange and circulatory efficiency. Circulation. 1996 Aug 15;94(4):842-7. doi: 10.1161/01.cir.94.4.842. PMID 8772709
- [Background] Schmidt M, Demoule A, Cracco C, Gharbi A, Fiamma MN, Straus C, Duguet A, Gottfried SB, Similowski T. Neurally adjusted ventilatory assist increases respiratory variability and complexity in acute respiratory failure. Anesthesiology. 2010 Mar;112(3):670-81. doi: 10.1097/ALN.0b013e3181cea375. PMID 20179505
- [Background] Guzzetti S, Borroni E, Garbelli PE, Ceriani E, Della Bella P, Montano N, Cogliati C, Somers VK, Malliani A, Porta A. Symbolic dynamics of heart rate variability: a probe to investigate cardiac autonomic modulation. Circulation. 2005 Jul 26;112(4):465-70. doi: 10.1161/CIRCULATIONAHA.104.518449. Epub 2005 Jul 18. PMID 16027252